CLINICAL TRIAL: NCT04258995
Title: A PHASE 2, OPEN-LABEL TRIAL TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A BOOSTER DOSE OF A GROUP B STREPTOCOCCUS 6 VALENT POLYSACCHARIDE CONJUGATE VACCINE (GBS6) IN HEALTHY ADULTS
Brief Title: A TRIAL TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A BOOSTER DOSE OF A GROUP B STREPTOCOCCUS 6 VALENT POLYSACCHARIDE CONJUGATE VACCINE (GBS6) IN HEALTHY ADULTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C1091007
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Results first posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Group B Streptococcal Infections
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Intervention Model Description: There are two arms in the study however based on the prior formulation received participants can only be enrolled into one predetermined arm in the study. Participants are assigned by an interactive response technology (IRT) based on prior formulation received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GBS6 no aluminum phosphate (GBS6 no AlPO4) (Experimental)
  Interventions: Biological: Group B streptoccous 6-valent polysaccharide conjugate vaccine (GBS6)
- GBS6 with aluminum phosphate (GBS6 with AlPO4) (Experimental)
  Interventions: Biological: Group B streptoccous 6-valent polysaccharide conjugate vaccine (GBS6)

INTERVENTIONS:
Biological: Group B streptoccous 6-valent polysaccharide conjugate vaccine (GBS6) — 2 formulations at 1 dose level
  Other Names: GBS6

SUMMARY:
This study is an extension to the completed first-in-human C1091001 study (NCT03170609) and is to evaluate the safety and immunogenicity of a single booster vaccine dose of GBS6, administered approximately 2 years or more after a primary GBS6 dose, to healthy adult males and nonpregnant women. The study will determine whether individuals who received a primary dose of GBS6 have additional benefit following a booster dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults (male and female) at enrollment who are determined by medical history, physical examination, and clinical judgment of the investigator to be eligible for inclusion in the study.
2. Participants who were enrolled in the C1091001 study, received GBS6, and completed the 1-month blood draw.

Exclusion Criteria:

1. Pregnant female participants; breastfeeding female participants; positive urine pregnancy test for women of childbearing potential (WOCBP) at Visit 1 (prior to vaccination); and WOCBP who are, in the opinion of the investigator, sexually active and at risk for pregnancy and fertile men and WOCBP who are unwilling or unable to use effective methods of contraception as outlined in this protocol from the signing of the informed consent until at least 3 months after the last dose of investigational product.
2. Acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study. Chronic medical conditions include human immunodeficiency virus, chronic hepatitis B virus (HBV) infection (HBV surface antigen positive), and/or hepatitis C virus infection.
3. History of severe adverse reaction and/or severe allergic reaction (eg, anaphylaxis) to any vaccine.
4. History of microbiologically proven invasive disease caused by group B streptococcus (Streptococcus agalactiae).
5. Previous vaccination with any licensed or investigational group B streptococcus vaccine (other than GBS6), or planned receipt during the participant's participation in the study (through 6-month telephone call).

Ages: 20 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Kentucky Pediatric & Adult Research Inc., Bardstown, Kentucky
  - J. Lewis Research, Inc./ Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Jongihlati B, Segall N, Block SL, Absalon J, Perez J, Munson S, Sanchez-Pearson Y, Simon R, Silmon de Monerri NC, Radley D, McLaughlin LC, Gaylord M, Gruber WC, Jansen KU, Scott DA, Anderson AS. Safety and immunogenicity of a booster dose of a novel hexavalent group B streptococcus conjugate vaccine in healthy, non-pregnant adults: a phase 2, open-label extension of a phase 1/2 randomised controlled trial. Lancet Infect Dis. 2025 Oct;25(10):1138-1148. doi: 10.1016/S1473-3099(25)00216-6. Epub 2025 Jun 13. PMID 40523378
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1091007

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, a total of 151 participants were assigned and vaccinated with a single booster dose of group B streptococcus 6-valent polysaccharide conjugate vaccine (GBS6) (20 microgram [μg] capsular polysaccharide [CPS]/serotype/dose) formulated with or without aluminum phosphate (AlPO4) based on the formulation received in the primary C1091001 study.
Groups:
- GBS6 20 μg With AlPO4: Participants who received a primary dose of GBS6 (5 μg, 10 µg, or 20 µg) with AlPO4 in Study C1091001 received a single booster dose of GBS6 (20 µg) formulated with AlPO4 intramuscularly on Day 1 and were followed up to 6 months.
- GBS6 20 μg Without AlPO4: Participants who received a primary dose of GBS6 (5 μg, 10 µg, or 20 µg) without AlPO4 in Study C1091001 received a single booster dose of GBS6 (20 µg) formulated without AlPO4 intramuscularly on Day 1 and were followed up to 6 months.
Period: Overall Study
Arm/Group | GBS6 20 μg With AlPO4 | GBS6 20 μg Without AlPO4
Started | 76 | 75
Vaccinated | 76 | 75
Completed | 75 | 74
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received 1 booster dose and had at least 1 safety assessment after receiving the booster dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | GBS6 20 μg With AlPO4 | GBS6 20 μg Without AlPO4 | Total
Number analyzed (Participants) | 76 | 75 | 151
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.1 (8.40) | 36.2 (8.96) | 36.7 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 60 | 114
  Male | 22 | 15 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 72 | 69 | 141
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 14 | 20
  White | 66 | 59 | 125
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Prompted Local Reactions Within 14 Days Following Booster Dose (Redness, Swelling, and Pain at the Injection Site)
Description: Local reactions were collected by using an e-diary and included pain at injection site, redness, and swelling graded below: pain at injection site: mild (did not interfere with activity), moderate (repeated use of nonnarcotic pain reliever >24 hours or interfered with activity), severe (any use of narcotic pain reliever or prevented daily activity), grade 4 (emergency room visit or hospitalization). Redness and swelling were graded as: mild (2.0-5.0 centimeter [cm]), moderate (greater than [>] 5.0-10.0 cm),severe (>10.0 cm), grade 4 for redness (necrosis or exfoliative dermatitis) and grade 4 for swelling (necrosis).Maximum severity (highest grading) of each location reaction within 14 days of vaccination was derived.
Time Frame: Within 14 days after booster dose
Population: All the participants reporting "yes" or "no" for at least 1 day were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GBS6 20 μg With AlPO4 | GBS6 20 μg Without AlPO4
Number analyzed (Participants) | 76 | 75
Percentage of participants
  Pain at injection site: Any | 68.4 [56.7 to 78.6] | 42.7 [31.3 to 54.6]
  Pain at injection site: Mild | 53.9 [42.1 to 65.5] | 38.7 [27.6 to 50.6]
  Pain at injection site: Moderate | 11.8 [5.6 to 21.3] | 4.0 [0.8 to 11.2]
  Pain at injection site: Severe | 2.6 [0.3 to 9.2] | 0 [0.0 to 4.8]
  Pain at injection site: Grade 4 | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]
  Redness: Any | 3.9 [0.8 to 11.1] | 2.7 [0.3 to 9.3]
  Redness: Mild | 3.9 [0.8 to 11.1] | 2.7 [0.3 to 9.3]
  Redness: Moderate | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]
  Redness: Severe | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]
  Redness: Grade 4 | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]
  Swelling: Any | 2.6 [0.3 to 9.2] | 4.0 [0.8 to 11.2]
  Swelling: Mild | 2.6 [0.3 to 9.2] | 4.0 [0.8 to 11.2]
  Swelling: Moderate | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]
  Swelling: Severe | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]
  Swelling: Grade 4 | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]

2. Primary Outcome: Percentage of Participants Reporting Prompted Systemic Events Within 14 Days Following Booster Dose (Fever, Nausea/Vomiting, Diarrhea, Headache, Fatigue, Muscle Pain, and Joint Pain)
Description: Nausea/Vomiting:Mild:No interference with activity or 1-2 times in 24 hours;Moderate:Some interference with activity or>2 times in 24 hours;Severe:Prevented daily activity, required IV hydration.Diarrhea:Mild:2-3 loose stools in 24 hours;Moderate: 4-5 loose stools in 24 hours;Severe:>=6 loose stools in 24 hours.Headache:Mild:No interference with activity;Moderate:Repeated use of nonnarcotic pain reliever >24 hours or some interference with activity;Severe:Significant; any use of narcotic pain reliever or prevents daily activity.Fatigue:Mild:No interference with activity;Moderate: Some interference with activity;Severe: Significant; prevented daily activity.Muscle pain:Mild: No interference with activity;Moderate:Some interference with activity;Severe:Significant;prevented daily activity.Muscle/joint pain:Mild: No interference with activity;Moderate:Some interference with activity;Severe:Significant; prevented daily activity.Grade 4 for all AEs:Emergency visit or hospitalization.
Time Frame: Within 14 days after booster dose
Population: All the participants reporting "yes" or "no" for at least 1 day were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GBS6 20 μg With AlPO4 | GBS6 20 μg Without AlPO4
Number analyzed (Participants) | 76 | 75
percentage of participants
  Fever:>=38.0 degree C | 3.9 [0.8 to 11.1] | 1.3 [0.0 to 7.2]
  Fever: 38.0°C to 38.4°C | 1.3 [0.0 to 7.1] | 0 [0.0 to 4.8]
  Fever: >38.4°C to 38.9°C | 2.6 [0.3 to 9.2] | 1.3 [0.0 to 7.2]
  Fever: >38.9°C to 40.0°C | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]
  Fever: >40.0°C | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]
  Nausea/vomiting: Any | 7.9 [3.0 to 16.4] | 10.7 [4.7 to 19.9]
  Nausea/vomiting: Mild | 6.6 [2.2 to 14.7] | 5.3 [1.5 to 13.1]
  Nausea/vomiting: Moderate | 1.3 [0.0 to 7.1] | 5.3 [1.5 to 13.1]
  Nausea/vomiting: Severe | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]
  Nausea/vomiting: Grade 4 | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]
  Diarrhea: Any | 15.8 [8.4 to 26.0] | 16.0 [8.6 to 26.3]
  Diarrhea: Mild | 14.5 [7.5 to 24.4] | 10.7 [4.7 to 19.9]
  Diarrhea: Moderate | 1.3 [0.0 to 7.1] | 5.3 [1.5 to 13.1]
  Diarrhea: Severe | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]
  Diarrhea: Grade 4 | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]
  Headache: Any | 30.3 [20.2 to 41.9] | 41.3 [30.1 to 53.3]
  Headache: Mild | 21.1 [12.5 to 31.9] | 26.7 [17.1 to 38.1]
  Headache: Moderate | 9.2 [3.8 to 18.1] | 13.3 [6.6 to 23.2]
  Headache: Severe | 0 [0.0 to 4.7] | 1.3 [0.0 to 7.2]
  Headache: Grade 4 | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]
  Fatigue/tiredness: Any | 44.7 [33.3 to 56.6] | 30.7 [20.5 to 42.4]
  Fatigue/tiredness: Mild | 23.7 [14.7 to 34.8] | 20.0 [11.6 to 30.8]
  Fatigue/tiredness: Moderate | 19.7 [11.5 to 30.5] | 9.3 [3.8 to 18.3]
  Fatigue/tiredness: Severe | 1.3 [0.0 to 7.1] | 1.3 [0.0 to 7.2]
  Fatigue/tiredness: Grade 4 | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]
  Muscle pain: Any | 23.7 [14.7 to 34.8] | 17.3 [9.6 to 27.8]
  Muscle pain: Mild | 11.8 [5.6 to 21.3] | 14.7 [7.6 to 24.7]
  Muscle pain: Moderate | 9.2 [3.8 to 18.1] | 2.7 [0.3 to 9.3]
  Muscle pain: Severe | 2.6 [0.3 to 9.2] | 0 [0.0 to 4.8]
  Muscle pain: Grade 4 | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]
  Joint pain: Any | 11.8 [5.6 to 21.3] | 9.3 [3.8 to 18.3]
  Joint pain: Mild | 6.6 [2.2 to 14.7] | 6.7 [2.2 to 14.9]
  Joint pain: Moderate | 3.9 [0.8 to 11.1] | 2.7 [0.3 to 9.3]
  Joint pain: Severe | 1.3 [0.0 to 7.1] | 0 [0.0 to 4.8]
  Joint pain: Grade 4 | 0 [0.0 to 4.7] | 0 [0.0 to 4.8]

3. Primary Outcome: Percentage of Participants Reporting Adverse Events (AEs) Within 1 Month Following Booster Dose
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or that was considered to be an important medical event. AEs included both non-serious AEs and SAEs.
Time Frame: Within 1 month after booster dose
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GBS6 20 μg With AlPO4 | GBS6 20 μg Without AlPO4
Number analyzed (Participants) | 76 | 75
percentage of participants | 6.6 [2.2 to 14.7] | 12.0 [5.6 to 21.6]

4. Primary Outcome: Percentage of Participants Reporting Medically Attended Adverse Events (MAEs) Within 6 Months Following Booster Dose
Description: An AE was any untoward medical occurrence in a participant in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or that was considered to be an important medical event. An MAE was defined as a non serious AE (AE other than SAE) that resulted in an evaluation at a medical facility.
Time Frame: Within 6 months after booster dose
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GBS6 20 μg With AlPO4 | GBS6 20 μg Without AlPO4
Number analyzed (Participants) | 76 | 75
percentage of participants | 11.8 [5.6 to 21.3] | 9.3 [3.8 to 18.3]

5. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Within 6 Months After Booster Dose
Description: An AE was any untoward medical occurrence in a participant in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or that was considered to be an important medical event.
Time Frame: Within 6 months after booster dose
Population: Safety population included all participants who received the booster dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GBS6 20 μg With AlPO4 | GBS6 20 μg Without AlPO4
Number analyzed (Participants) | 76 | 75
percentage of participants | 1.3 [0.0 to 7.1] | 0 [0.0 to 4.8]

6. Secondary Outcome: GBS Serotype-Specific IgG Geometric Mean Concentrations (GMC) Measured Before and 1 Month After Booster Dose
Description: Serotypes used for evaluation were: Ia, Ib, II, III, IV, and V.
Time Frame: Before and 1 month after booster dose
Population: Evaluable immunogenicity population included participants who had received 1 booster dose (as assigned); had a Visit 2 blood draw within 27 to 45 days after booster dose administration; had at least 1 valid and determinate assay result at Visit 2; and had no major protocol violation.
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per milliliter
Arm/Group | GBS6 20 μg With AlPO4 | GBS6 20 μg Without AlPO4
Number analyzed (Participants) | 76 | 74
Microgram per milliliter
  Ia: Day 1 - Booster Dose | 3.070 [1.539 to 6.125] | 3.252 [1.558 to 6.787]
  Ia: Month 1 - Booster Dose | 47.600 [34.705 to 65.285] | 52.038 [35.654 to 75.951]
  Ib: Day 1 - Booster Dose | 0.537 [0.272 to 1.060] | 0.588 [0.302 to 1.146]
  Ib: Month 1 - Booster Dose | 24.298 [17.396 to 33.940] | 20.095 [14.033 to 28.775]
  II: Day 1 - Booster Dose | 5.244 [3.186 to 8.630] | 6.379 [4.007 to 10.155]
  II: Month 1 - Booster Dose | 51.670 [39.310 to 67.916] | 64.617 [47.313 to 88.249]
  III: Day 1 - Booster Dose | 0.850 [0.508 to 1.423] | 1.227 [0.750 to 2.008]
  III: Month 1 - Booster Dose | 13.511 [10.224 to 17.854] | 17.305 [12.994 to 23.046]
  IV: Day 1 - Booster Dose | 0.768 [0.496 to 1.189] | 0.873 [0.573 to 1.329]
  IV: Month 1 - Booster Dose | 30.048 [23.259 to 38.818] | 33.216 [24.452 to 45.120]
  V: Day 1 - Booster Dose | 1.104 [0.608 to 2.004] | 0.992 [0.556 to 1.771]
  V: Month 1 - Booster Dose | 39.368 [27.387 to 56.589] | 52.326 [36.887 to 74.227]

7. Secondary Outcome: GBS Serotype-Specific Opsonophagocytic Activity (OPA) Geometric Mean Titers Measured Before to 1 Month After Booster Dose
Description: OPA for the 6 serotypes (Ia, Ib, II, III, IV, V) were determined in all participants for each blood sample at Day 1 and at 1 month after booster dose.
Time Frame: Within 6 months after primary dose and within 1 month after booster dose
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GBS6 20 μg With AlPO4 | GBS6 20 μg Without AlPO4
Number analyzed (Participants) | 76 | 74
Titer
  Ia: Day 1 - Booster Dose: number analyzed (Participants) | 74 | 74
  Ia: Day 1 - Booster Dose | 1368 [826 to 2266] | 1361 [831 to 2228]
  Ia: Month 1 - Booster Dose | 9374 [7164 to 12266] | 8809 [6665 to 11643]
  Ib: Day 1 - Booster Dose: number analyzed (Participants) | 75 | 71
  Ib: Day 1 - Booster Dose | 3307 [1993 to 5487] | 2734 [1603 to 4662]
  Ib: Month 1 - Booster Dose: number analyzed (Participants) | 75 | 74
  Ib: Month 1 - Booster Dose | 28809 [21345 to 38883] | 18550 [12943 to 26586]
  II: Day 1 - Booster Dose | 3209 [2266 to 4545] | 3659 [2705 to 4950]
  II: Month 1 - Booster Dose: number analyzed (Participants) | 75 | 74
  II: Month 1 - Booster Dose | 16057 [12486 to 20650] | 15317 [11689 to 20071]
  III: Day 1 - Booster Dose: number analyzed (Participants) | 74 | 74
  III: Day 1 - Booster Dose | 756 [508 to 1126] | 641 [432 to 951]
  III: Month 1 - Booster Dose | 3695 [2776 to 4917] | 3339 [2381 to 4681]
  IV: Day 1 - Booster Dose | 5591 [4295 to 7279] | 4617 [3429 to 6217]
  IV: Month 1 - Booster Dose | 22994 [18192 to 29063] | 19710 [15517 to 25035]
  V: Day 1 - Booster Dose | 2249 [1498 to 3376] | 2324 [1517 to 3560]
  V: Month 1 - Booster Dose | 10484 [7993 to 13750] | 8802 [6417 to 12073]

8. Secondary Outcome: GBS Serotype-Specific IgG Geometric Mean Fold Rise (GMFR) From Before To 1 Month After Booster Dose
Description: IgG for the 6 serotypes (Ia, Ib, II, III, IV, V) were determined in all participants for each blood sample at Day 1 and at 1 month after booster dose.
Time Frame: 1 month after booster dose
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | GBS6 20 μg With AlPO4 | GBS6 20 μg Without AlPO4
Number analyzed (Participants) | 76 | 74
Fold rise
  Ia: Month 1 - Booster Dose | 15.504 [9.452 to 25.430] | 16.003 [9.800 to 26.132]
  Ib: Month 1 - Booster Dose | 45.282 [27.919 to 73.441] | 34.191 [21.272 to 54.955]
  II: Month 1 - Booster Dose | 9.853 [6.783 to 14.313] | 10.130 [6.822 to 15.042]
  III: Month 1 - Booster Dose | 15.889 [10.138 to 24.902] | 14.100 [9.453 to 21.031]
  IV: Month 1 - Booster Dose | 39.133 [26.569 to 57.638] | 38.063 [26.189 to 55.321]
  V: Month 1 - Booster Dose | 35.668 [23.796 to 53.463] | 52.750 [34.308 to 81.107]

9. Secondary Outcome: GBS Serotype-Specific OPA GMFR Measured Before and 1 Month After Booster Dose
Description: as for outcome 7
Time Frame: 1 month after booster dose
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | GBS6 20 μg With AlPO4 | GBS6 20 μg Without AlPO4
Number analyzed (Participants) | 76 | 74
Fold rise
  Ia: Month 1 - Booster Dose: number analyzed (Participants) | 74 | 74
  Ia: Month 1 - Booster Dose | 6.9 [4.80 to 10.00] | 6.5 [4.43 to 9.45]
  Ib: Month 1 - Booster Dose: number analyzed (Participants) | 74 | 71
  Ib: Month 1 - Booster Dose | 9.1 [6.21 to 13.47] | 6.4 [4.46 to 9.30]
  II: Month 1 - Booster Dose: number analyzed (Participants) | 75 | 74
  II: Month 1 - Booster Dose | 4.8 [3.65 to 6.36] | 4.2 [3.08 to 5.68]
  III: Month 1 - Booster Dose: number analyzed (Participants) | 74 | 74
  III: Month 1 - Booster Dose | 4.8 [3.54 to 6.58] | 5.2 [3.79 to 7.15]
  IV: Month 1 - Booster Dose | 4.1 [3.18 to 5.32] | 4.3 [3.17 to 5.74]
  V: Month 1 - Booster Dose | 4.7 [3.27 to 6.65] | 3.8 [2.63 to 5.45]

10. Secondary Outcome: GBS Serotype-Specific IgG GMC Measured 1 Month After Booster Dose Stratified by Baseline Pre-vaccination Status (Before the Primary Dose)
Description: Serotypes used for evaluation were: Ia, Ib, II, III, IV, and V. The pre-vaccination immunogenicity blood draw and booster vaccination were both performed on Day 1.
Time Frame: 1 month after booster dose
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter
Arm/Group | GBS6 20 μg With AlPO4 | GBS6 20 μg Without AlPO4
Number analyzed (Participants) | 76 | 74
microgram per milliliter
  Ia: Month 1 - Booster Dose Month 1 - Booster Dose = Positive: number analyzed (Participants) | 2 | 8
  Ia: Month 1 - Booster Dose Month 1 - Booster Dose = Positive | 55.766 [0.000 to 30690052.300] | 148.088 [50.544 to 433.884]
  Ia: Month 1 - Booster Dose Month 1 - Booster Dose = Negative: number analyzed (Participants) | 74 | 66
  Ia: Month 1 - Booster Dose Month 1 - Booster Dose = Negative | 47.396 [34.343 to 65.412] | 45.843 [30.695 to 68.465]
  Ib: Month 1 - Booster Dose Month 1 - Booster Dose = Positive: number analyzed (Participants) | 4 | 2
  Ib: Month 1 - Booster Dose Month 1 - Booster Dose = Positive | 40.327 [3.968 to 409.881] | 112.434 [0.000 to 245914635.435]
  Ib: Month 1 - Booster Dose Month 1 - Booster Dose = Negative: number analyzed (Participants) | 72 | 72
  Ib: Month 1 - Booster Dose Month 1 - Booster Dose = Negative | 23.624 [16.732 to 33.353] | 19.156 [13.365 to 27.456]
  II: Month 1 - Booster Dose Month 1 - Booster Dose = Positive: number analyzed (Participants) | 7 | 9
  II: Month 1 - Booster Dose Month 1 - Booster Dose = Positive | 189.611 [105.577 to 340.534] | 52.439 [18.337 to 149.961]
  II: Month 1 - Booster Dose Month 1 - Booster Dose = Negative: number analyzed (Participants) | 69 | 65
  II: Month 1 - Booster Dose Month 1 - Booster Dose = Negative | 45.285 [34.250 to 59.876] | 66.513 [47.596 to 92.948]
  III: Month 1 - Booster Dose Month 1 - Booster Dose = Positive: number analyzed (Participants) | 3 | 6
  III: Month 1 - Booster Dose Month 1 - Booster Dose = Positive | 22.612 [4.268 to 119.786] | 18.368 [6.559 to 51.438]
  III: Month 1 - Booster Dose Month 1 - Booster Dose = Negative: number analyzed (Participants) | 73 | 68
  III: Month 1 - Booster Dose Month 1 - Booster Dose = Negative | 13.228 [9.915 to 17.647] | 17.214 [12.681 to 23.366]
  IV: Month 1 - Booster Dose Month 1 - Booster Dose = Positive: number analyzed (Participants) | 2 | 3
  IV: Month 1 - Booster Dose Month 1 - Booster Dose = Positive | 48.545 [0.000 to 347896565796] | 77.627 [22.933 to 262.759]
  IV: Month 1 - Booster Dose Month 1 - Booster Dose = Negative: number analyzed (Participants) | 74 | 71
  IV: Month 1 - Booster Dose Month 1 - Booster Dose = Negative | 29.661 [23.021 to 38.216] | 32.046 [23.360 to 43.960]
  V: Month 1 - Booster Dose Month 1 - Booster Dose = Positive: number analyzed (Participants) | 4 | 1
  V: Month 1 - Booster Dose Month 1 - Booster Dose = Positive | 96.017 [19.528 to 472.109] | 103.130
  V: Month 1 - Booster Dose Month 1 - Booster Dose = Negative: number analyzed (Participants) | 72 | 73
  V: Month 1 - Booster Dose Month 1 - Booster Dose = Negative | 37.465 [25.698 to 54.622] | 51.842 [36.385 to 73.865]

ADVERSE EVENTS:
Time Frame: The time period for actively eliciting and collecting AEs and SAEs for each participant began from the time the participant provided informed consent, through and including Visit 2 (1 month after booster dose) for AEs and through and including Visit 3 for MAEs and SAEs (6 months after booster dose).
Description: Safety population are participants who received 1 dose of the investigational product and had at least 1 safety assessment after receiving the booster dose. Medical Dictionary for Regulatory Activities (MedDRA) v23.1 was followed for AE reporting.
Arm/Group | GBS6 20 μg With AlPO4 | GBS6 20 μg Without AlPO4
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/75
Serious Adverse Events (participants affected / at risk) | 1/76 | 0/75
Other Adverse Events (participants affected / at risk) | 59/76 | 54/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GBS6 20 μg With AlPO4 (N=76) | GBS6 20 μg Without AlPO4 (N=75)
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GBS6 20 μg With AlPO4 (N=76) | GBS6 20 μg Without AlPO4 (N=75)
Diarrhoea (Gastrointestinal disorders) | 12 | 12
Vomiting (Gastrointestinal disorders) | 6 | 8
Fatigue (General disorders) | 34 | 23
Injection site pain (General disorders) | 52 | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 13
Headache (Nervous system disorders) | 23 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT04258995/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT04258995/SAP_001.pdf